CLINICAL TRIAL: NCT03284814
Title: Single-dose and Multiple-dose Comparative Bioavailability Study of Three CoQ10 Formulations in Healthy Elderly Adults
Brief Title: Bioavailability Study of CoQ10 Formulations in Healthy Elderly Adults
Acronym: CoQ10-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Vizera d.o.o. (Industry); Valens Int. d.o.o., Slovenija (Industry); MEDEDUS, Ljubljana, Slovenia (Unknown)
Responsible Party: Principal Investigator, Snežana Kocijančič, PhD, Institute of Nutrition, Slovenia (Nutris)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KME 89/07/17
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Bioavailability of Coenzyme Q10
Keywords: coenzyme q10; single dose bioavailability; multiple dose bioavailability
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Three-period crossover bioavailability study will include 21 subjects who will test three CoQ10 formulations. Subjects will test 3 formulations of single dose CoQ10 within first 3 weeks to assess bioavailability, which will be followed with 2 weeks of continuous administration of one of study formulations to demonstrate and assesse multiple-dose profile of CoQ10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard product group (Active Comparator): This group will be included in a single dose cross over study, and in multiple dose study with standard product (SP: CoQ10 hard capsules; 100 mg)
  Interventions: Dietary Supplement: Single dose intervention with Standard product (SP); Dietary Supplement: Single dose intervention with Comparative product (CP); Dietary Supplement: Single dose intervention with Investigational product (IP); Dietary Supplement: Multiple dose intervention with Standard product (SP)
- Comparative product group (Active Comparator): This group will be included in a single dose cross over study, and in multiple dose study with comparative product (CP: CoQ10 soft-gel capsules; 100 mg)
  Interventions: Dietary Supplement: Single dose intervention with Standard product (SP); Dietary Supplement: Single dose intervention with Comparative product (CP); Dietary Supplement: Single dose intervention with Investigational product (IP); Dietary Supplement: Multiple dose intervention with Comparative product (CP)
- Investigational product group (Experimental): This group will be included in a single dose cross over study, and in multiple dose study with investigational product (IP: CoQ10 syrup; 100 mg)
  Interventions: Dietary Supplement: Single dose intervention with Standard product (SP); Dietary Supplement: Single dose intervention with Comparative product (CP); Dietary Supplement: Multiple dose intervention with Investigational product (IP)

INTERVENTIONS:
Dietary Supplement: Single dose intervention with Standard product (SP) — hard capsules, 100 mg
Dietary Supplement: Single dose intervention with Comparative product (CP) — soft-gel capsules, 100 mg
Dietary Supplement: Single dose intervention with Investigational product (IP) — syrup, 100 mg
  Arms: Comparative product group; Standard product group
Dietary Supplement: Multiple dose intervention with Standard product (SP) — hard capsules, 100 mg - 14 days
  Arms: Standard product group
Dietary Supplement: Multiple dose intervention with Comparative product (CP) — soft-gel capsules, 100 mg - 14 days
  Arms: Comparative product group
Dietary Supplement: Multiple dose intervention with Investigational product (IP) — syrup, 100 mg - 14 days
  Arms: Investigational product group

SUMMARY:
The single-center, randomized, open-label, three-period crossover bioavailability study will include 21 subjects who will test three CoQ10 formulations. Subjects will test 3 formulations of single dose CoQ10 within first 3 weeks to assess bioavailability, which will be followed with 2 weeks of continuous administration of one of study formulations to demonstrate and assesse multiple-dose profile of CoQ10.

ELIGIBILITY:
Inclusion Criteria:

* Subject Informed consent form (ICF) is singed
* Aged between 65 and 74 years at the time of the signature of ICF
* A body mass index between 20 and 29 kg/m2
* Healthy, meaning absence of any prescribed medication for a month prior to the inclusion to the study and during the study
* Willing to avoid a consumption of any food supplements except vitamin D and calcium at least 2 weeks before and during the study
* Consumption of dairy and cereal products (standardised breakfast will include low lactose dairy and bread)
* Willing to follow all study procedures, including attending all site visits (including sessions during which a venous line will be inserted for blood sampling), and keeping a diary for the time of multiple-dose study (to follow their compliance and palatability)

Exclusion Criteria:

* Intake of any prescribed medication within 2 weeks of the beginning of the study
* Intake of any food supplements within 2 weeks of the beginning of the study, except vitamin D and calcium
* Hypotension
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular or hematological disease, diabetes
* Gastrointestinal disorders or other serious acute or chronic diseases
* Known lactose/gluten intolerances/ food allergies (limitation for standardisation of meals)
* Inadequate veins (in the opinion of the investigator) or known contraindication to placement of a dedicated peripheral line for venous blood withdrawal
* Known drug and/or alcohol abuse
* Using any form of nicotine or tobacco
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another investigational study or blood donation within 3 months prior to or during this study

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
improved single dose bioavailability of IP (in comparison to SP) | 48 hours
  Relative bioavailability between the investigational and standard product expressed as ratio of AUC0-48h (area under the plasma concentration curve from the administration time to the last observation point, i.e. 48h) of total CoQ10 plasma concentrations above the baseline value.
improved plasma CoQ10 level after multiple dose study for IP (in comparison to SP) | 14 days
  Ratio between total CoQ10 trough plasma concentrations after multiple-dose application on day 14 (CMIN,day14) between the investigational and standard product.

SECONDARY OUTCOMES:
comparable single dose bioavailability of IP (in comparison to CP) | 48 hours
  Relative bioavailability between the investigational product and comparator expressed as ratio of AUC0-48h of total CoQ10 plasma concentrations above the baseline value.
comparable plasma CoQ10 level after multiple dose study for IP (in comparison to CP) | 14 days
  Ratio between total CoQ10 trough plasma concentrations after multiple-dose application on day 14 (CMIN,day14) between the investigational product and comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, Principal Investigator — Nutrition Institute, Ljubljana; Snežana Kocijančič, Principal Investigator — MEDEDUS, Ljubljana, Slovenia
Locations (3):
- Slovenia (3):
  - MEDEDUS, Ljubljana, Slovenia, Ljubljana
  - Nutrition Institute, Ljubljana, Ljubljana
  - Vizera d.o.o., Ljubljana, Slovenia, Ljubljana